CLINICAL TRIAL: NCT04176172
Title: Testing Novel Pharmacogenetic and Adherence Optimization Treatments to Improve the Effectiveness of Smoking Cessation Treatments for Smokers With HIV
Brief Title: Optimizing Tobacco Use Treatment for PLWHA
Acronym: HTO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Northwestern University (Other)
Responsible Party: Principal Investigator, Robert Schnoll, Professor and Director, Center for Interdisciplinary Research on Nicotine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 834345; 1R01CA243914-01 (NIH)
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: HIV/AIDS; Nicotine Dependence
Keywords: Smoking Cessation; Nicotine Dependence; HIV/AIDS; Varenicline; Nicotine Patch; Cigarette Smoking; Managed Problem Solving
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tobacco Use Disorder; Smoking Cessation; Cigarette Smoking | interventions — Varenicline; Tobacco Use Cessation Devices; Nicotine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Varenicline & Standard Cessation Counseling (Active Comparator): varenicline plus standard behavioral smoking cessation treatment
  Interventions: Drug: Varenicline; Behavioral: Standard treatment
- NMR-Tailored Medication & Standard Cessation Counseling + MAPS (Experimental): varenicline or nicotine patch plus standard behavioral smoking cessation treatment with Managed Problem Solving adherence intervention
  Interventions: Drug: Varenicline; Drug: Nicotine patch; Behavioral: Standard treatment + Managed Problem Solving (MAPS) adherence intervention

INTERVENTIONS:
Drug: Varenicline — Participants will receive open-label varenicline for 12 weeks.
  Other Names: Chantix or Apo-Varenicline
Drug: Nicotine patch — Participants will receive open-label nicotine patch for 12 weeks. (Participants in the NMR-tailored treatment arms will receive either varenicline OR patch; they will not receive both)
  Other Names: NicoDerm
  Arms: NMR-Tailored Medication & Standard Cessation Counseling + MAPS
Behavioral: Standard treatment — Standard behavioral smoking cessation treatment is an effective treatment for nicotine dependence. Treatment focuses on self-monitoring of smoking behavior, identifying smoking triggers and alternative trigger management strategies, relaxation, social support for non-smoking, and relapse prevention. Participants will receive up to 5 therapy sessions (2 in person, 3 over the phone) over 8 weeks.
  Other Names: Standard Therapy
  Arms: Varenicline & Standard Cessation Counseling
Behavioral: Standard treatment + Managed Problem Solving (MAPS) adherence intervention — Standard behavioral smoking cessation treatment is an effective treatment for nicotine dependence. Treatment focuses on self-monitoring of smoking behavior, identifying smoking triggers and alternative trigger management strategies, relaxation, social support for non-smoking, and relapse prevention. Managed Problem Solving (MAPS) is a therapeutic process that involves the systematic delineation of a participant's medication adherence problems and construction of a series of individualized solutions that therapists and participants explore together. Participants will receive up to 5 therapy sessions (2 in person, 3 over the phone) over 8 weeks. The first session will directly address potential medication adherence barriers, and therapist and participant will collaboratively brainstorm ways to overcome these barriers.
  Other Names: Standard treatment + MAPS
  Arms: NMR-Tailored Medication & Standard Cessation Counseling + MAPS

SUMMARY:
The advent of anti-retroviral therapy (ART) for people living with HIV/AIDS (PLWHA) substantially improved life expectancy but has also led to the critical need to address modifiable risk factors associated with cancer and cardiovascular disease, such as tobacco smoking. HIV-infected smokers lose more life-years due to tobacco use than they do to their HIV infection.

There have been relatively few studies of tobacco use treatments for PLWHA and systematic reviews show that there are insufficient data to conclude that tobacco dependence interventions that are efficacious in the general population are efficacious for PLWHA. Further, many studies in this area have lacked randomization and a control group, infrequently used an intent-to-treat (ITT) approach and biological verification of tobacco abstinence, and lacked post-treatment follow-up.10 What investigators do know thus far is that behavioral interventions and the nicotine patch yield moderate effects on cessation; and 2 recent placebo-controlled trials - one in France and one by this lab - found that varenicline is safe and effective for treating tobacco use among PLWHA, but yield quit rates that are substantially lower than those reported in the general population. Thus, there is a critical need to rigorously test novel ways to optimize tobacco cessation treatment for smokers with HIV.

DETAILED DESCRIPTION:
Smoking among PLWHA is a critical public health issue, with the rate of smoking 2-3 times greater than it is in the general population and the health risks of smoking outweighing those associated with the virus itself. Unfortunately, remarkably few studies have evaluated smoking cessation interventions for PLWHA and the available literature indicates that both behavioral and pharmacological smoking cessation interventions yield modest effect sizes and quit rates that are considerably lower than in the general population. A sizable literature, including studies by our research team, indicates that using the nicotine metabolite ratio (NMR) to personalize the selection of medications for tobacco use and the MAPS intervention to augment adherence to these medications can optimize treatments for tobacco use among PLWHA. The NCI recognized the potential for clinicians to use the NMR to individualize cessation treatment in order to improve effectiveness (https://www.cancer.gov/about-nci/budget/plan/public-health) and the Centers for Disease Control and Prevention (CDC) has endorsed MAPS as an evidence-based approach to increasing medication adherence among PLWHA. As such, this trial will test these intervention optimization strategies to determine if individually or together they can represent an effective approach to treating tobacco use in this under-served population of smokers. As a major advance for this area of work, the investigators will use rigorous methodology to evaluate these optimization strategies (i.e., a randomized design, biological verification, an ITT approach, and 6-month outcome assessments) and, overall, our approach is consistent with the multiphase optimization strategy (MOST) framework, which has been used to identify intervention components that maximize cessation outcomes. This trial will also assess theoretically derived and empirically based mechanisms through which these optimization strategies affect cessation and explore sub-groups who are more or less responsive to these strategies. In the end, this trial, which is consistent with the Office of AIDS Research trans-NIH Strategic Plan for HIV and HIV-Related Research (https://www.oar.nih.gov/hiv-policy-and-research/research-priorities), will determine if getting the right medication to the right person and making sure they adequately use the medication optimizes tobacco cessation treatments among PLWHA as a critical way to improve health outcomes for this population.

ELIGIBILITY:
Key Inclusion Criteria:

* >18 years, smoke daily for the past 30 days
* Confirmed HIV+ (exhibit viral load of <1000 copies/mL)
* Residing in the geographic area close to one of the sites for at least 7 months
* Able to use varenicline/TN patch safely

Key Exclusion Criteria:

* Current untreated and unstable diagnosis of substance abuse/dependence
* Current diagnosis of unstable and untreated major depression, psychosis or bipolar disorder
* Suicide risk as measured by the C-SSRS
* Current use or discontinuation within last 14 days of quit smoking medications
* Cancer, heart disease, stroke or MI within the past 6 months requires study physician approval
* Uncontrolled hypertension
* History of epilepsy or seizure disorder requires study physician approval
* Women who are pregnant, planning a pregnancy, or lactating
* Use of e-cigarettes, chewing tobacco, snuff or snus
* Generalized eczema or psoriasis
* A reaction or sensitivity to a nicotine patch or any other transdermal medication requires study physician approval
* Currently participating in a smoking cessation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Point-prevalence abstinence | 26 weeks (24 weeks post target quit date)
  Participants will be considered abstinent if they report abstinence, not even a puff of a cigarette, for >7 days prior to week 26 (24 weeks post target quit date) and have an expired carbon monoxide reading of ≤8 parts per million at week 26.

SECONDARY OUTCOMES:
Six-month quit rate | 6 months
  The number of days in a six-month period of self-reported smoking
Prolonged abstinence | 26 weeks (24 weeks post target quit date)
  <7 consecutive days of self-reported smoking after a 2-week grace period
Continuous abstinence | 26 weeks (24 weeks post target quit date)
  No smoking between target quit date (week 2) and week 26
Time to 7-day relapse | 26 weeks (24 weeks post target quit date)
  Time to relapse as defined by 7 or more consecutive days of self-reported smoking (no grace period)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schnoll, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania